CLINICAL TRIAL: NCT01618682
Title: Cortical Organization in Allogeneic Transplants or Heterotopic Hand Replants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 11.0616
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Hand Transplant; Hand Replant
Keywords: hand transplant; hand replant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hand Transplant Patients: These will be subjects who have undergone a hand transplant.
- Hand Replant Patients: These will be patients who have undergone a hand replant procedure.

SUMMARY:
The investigators hope to gain insights into the functional organization of the human cerebral cortex in response to upper limb amputation and surgical interventions including hand replantation and hand transplantation.

ELIGIBILITY:
Inclusion Criteria:

* between 18-70 yrs old
* undergone successful allogeneic transplantation of one or both hands OR undergone successful reattachment of one or both hands OR will have experienced surgical repair of one or more severed nerves (ulnar, medial, radial, digital in the upper limb
* must speak English

Exclusion Criteria:

* younger than 18 years or older than 70 years
* not undergone a replant or transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be patients who have undergone hand transplant or replant procedures at Kleinert Kutz and Associates or who are on the hand transplant registry.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Biomicroscopy | Up to 12 months
  We will scan the cross section of the medial nerve at the pisiform bone level to determine the level of CTS with Ultrasound Biomicroscopy machine. This device is not approved for clinical decisions, only used for research purposes.

SECONDARY OUTCOMES:
Grip Strength | Up to 12 months
Pinch Strength | Up to 12 months
DASH Questionnaire | Up to 12 months
  Subjects will complete the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Kaufman, PhD, Principal Investigator — Christine M. Kleinert Institute for Hand and Microsurgery
Locations (1):
- Christine M. Kleinert Insitute of Hand and Microsurgery, Louisville, Kentucky, United States